CLINICAL TRIAL: NCT02567357
Title: PREDICTORS (Parents Resources for Decreasing the Incidence of Change Triggered Temper Outbursts)
Brief Title: Parents Resources for Decreasing the Incidence of Change Triggered Temper Outbursts
Acronym: PREDICTORS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: University of Warwick (Other); University of Birmingham (Other)
Responsible Party: Principal Investigator, Kate Woodcock, Lecturer, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R2149PSY
Record Dates: First submitted 2015-09-24; First posted 2015-10-05 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2016-09

CONDITIONS: Child Behavior
Keywords: change triggered temper outbursts; parent training; autism; intellectual disability; Prader-Willi syndrome; Fragile X syndrome; web-based training; Down syndrome
MeSH Terms: conditions — Child Behavior; Autistic Disorder; Intellectual Disability; Prader-Willi Syndrome; Fragile X Syndrome; Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visual Scheduling (Active Comparator): A caregiver training package on the use of a pictorial (visual) schedule to illustrate each day's expected activities to a child. Caregivers will be trained to ensure that activities occur as described in the schedule as far as possible, thus the expected mechanism of action is the reduction of (unexpected change) antecedents of children's temper outbursts.
  Interventions: Behavioral: Visual Scheduling
- Signalling change (Experimental): A caregiver training package where parents are taught to present a distinctive visual-verbal cue to a child whenever they become aware that a change will take place in the child's usual/expected activities. Caregivers will be trained to only ever present to cue if they can be sure that a change to the child's routine or plan will occur, thus the expected mechanism of action is the child's learned association between the presentation of the cue and the subsequent occurrence of a change to their expectations. Signalled changes will therefore be more predictable for the child, and should therefore be easier for them to deal with.
  Interventions: Behavioral: signalling change

INTERVENTIONS:
Behavioral: Visual Scheduling — Caregivers will present a visual schedule with pictorial representations of activities/events expected to occur each day will be presented to children at set times of day (tailored for individual's schedules). Ultimately caregivers will aim to ensure that activities occur as per the schedule as far as possible - thus decreasing the child's level of exposure to unexpected changes in routines or plans.
  Other Names: antecedent manipulation
  Arms: Visual Scheduling
Behavioral: signalling change — Caregivers will present a distinct visual-verbal cue card whenever they become aware that a change to the child's routine or plan is about to occur. Thus, the intervention uses a stimulus control approach so that the child learns that presentation of the cue reliably predicts the subsequent occurrence of a change to routine/plan, and the change is therefore more predictable and easier for the child to deal with.
  Other Names: cuing change
  Arms: Signalling change

SUMMARY:
'PREDICTORS' (Parents Resources for Decreasing the Incidence of Change Triggered Temper Outbursts) aims to evaluate web-based training packages for caregivers of children who show frequent temper outbursts following changes to their routines and plans. The training packages will teach caregivers how to apply strategies that aim to reduce the number of temper outbursts that the children show following changes, as well as making any outbursts they do show less severe (less functionally impairing).

DETAILED DESCRIPTION:
The aims of PREDICTORS are: 1. To refine the tools to implement and evaluate a resource-efficient caregiver training program for signalling changes to children with intellectual disabilities or autism spectrum disorders. 2. To pilot the program to test the feasibility of taking it forward into a clinical trial. 3. To conduct a process and economic evaluation of the pilot intervention to provide further data on its suitability for a clinical trial.

Parents/caregivers of children aged 7-16 years old who frequently show temper outbursts when things change in their routines or plans will keep a web-based diary accessed via smart phone or other device on their child's temper outbursts for a 6 month period (baseline). After 6 months of keeping this diary, parents/caregivers will then access web-based training for approximately 1 month which will include sessions to study once or twice per week as well as exercises to practice in between sessions.

After the training is complete parents will be asked to implement the strategies they have learnt in the 6 months that follow. In addition researchers from the university will telephone parents/ caregivers to ask some questions about their child's temper outbursts and on the effects this behaviour has on daily life. Parents will be interviewed at three points during the study (before baseline, after baseline, before intervention and after intervention phases). Interviews will focus on gathering information of their child's behaviour.

Focus groups with relevant experienced professionals and parents (not participating in the main part of the study) will guide the training resource development and development and content of the behaviour diary used by parents during the study.

ELIGIBILITY:
Inclusion Criteria:

* children aged 7-16 years of age, with temper outbursts triggered by change to routine or plans and their parent(s)/caregiver(s)

Exclusion Criteria:

* children who show less than one change triggered temper outburst (temper outbursts following an unexpected change in plan, routine or expectation) per month

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in frequency of temper outbursts between baseline and intervention | 6 months baseline, 6 months during intervention
  Informant reports of outbursts using a web-based behaviour diary after they occur. Entries comprise check lists of individual behaviours comprised in the outburst, an intensity rating (1-3 or 1-5 point scale depending on the different intensities of outburst parents were able to operationally describe), a description of the duration (<1 minute; >1 & <5 minutes; >5 & <15 minutes; >15 minutes & < 1 hour; >1 hour [specify]); a check list of possible antecedent events; and a check list of possible actions taken by caregivers. Frequency per month of temper outbursts following change-related antecedents of each intensity level and each duration will comprise the primary measurement.
  Reports will also be made every 3 days, of the number of outbursts over the previous 3 days (for validity checking); and of the number of changes to routines/plans experienced by the child. The percentage of changes that were followed by outbursts will comprise measurement 2.
Change in percentage of changes to routines/plans experienced by children that are followed by temper outbursts between baseline and intervention | 6 months baseline, 6 months during intervention
  Informant reports will be made using a scheduled entry section of the behaviour diary, on the number of changes to routines /plans experienced by the child since the previous entry. These data will be used to calculate the percentage of experienced changes that were followed by a temper outburst

SECONDARY OUTCOMES:
Change in cost of services with which the child engages - Cost of Services Receipt Inventory | within 2 weeks before baseline, within one month after baseline, within one month following intervention
  An informant report questionnaire on the cost to health services associated with the child over the previous 6 months
Process information on how the intervention strategies are being implemented by caregivers | every three days for 7 months from after baseline onwards
  Informant report ratings on the use of the intervention strategy and how easy this was

CONTACTS AND LOCATIONS:
Overall Officials: Kate Woodcock, PhD, Study Director — Queen's Univerisity Belfast
Locations (1):
- Queen's University Belfast, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Behaviour diary (primary outcome measure) can be viewed via test code 794613 — http://www.psych.qub.ac.uk/surveys/predictors/